CLINICAL TRIAL: NCT04864847
Title: A Study of Contrast-induced Acute Kidney Injury Prediction Using the RENISCHEM L-FABP Assay at the Point-of-Care
Brief Title: Clinical Validation of the RENISCHEM L-FABP POC Assay
Acronym: SAKURA-POC
Status: Recruiting | Type: Observational
Sponsor: Hikari Dx, Inc. (Other)
Collaborators: Timewell Medical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: TWM-001
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Acute Kidney Injury; Contrast-induced Nephropathy
Keywords: L-FABP; Point of Care
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: RENISCHEM L-FABP POC Test — Point-of-care test cassette with quantitative reader used for the measurement of L-type fatty acid binding protein (L-FABP) in human urine specimens.

SUMMARY:
This study will involve measurement of levels of a novel urinary biomarker of renal ischemia, L-FABP. The purpose of the study is to perform a clinical validation of the ability of L-FABP measurements in urine using the RENISCHEM L-FABP POC Test to predict the development of AKI within 2 days following cardiac and vascular catheterization procedures involving exposure to radiocontrast media.

DETAILED DESCRIPTION:
This study will validate the ability of the RENISCHEM L-FABP POC test to predict AKI risk in patients undergoing cardiac catheterization and receiving iodinated contrast medium. Contrast medium is known to be both vasoconstrictive and chemotoxic, which can lead to renal ischemia and, ultimately, AKI. Infusion of radiographic contrast agents, with the associated increases in osmotic load and viscosity, increases hypoxia of the renal medulla and increases renal free radical production through post-ischemic oxidative stress. Earlier identification of contrast medium-induced acute kidney injury (CI-AKI) risk can facilitate improved management of patients to prevent AKI, for example, through selection of alternative imaging methods or contrast agents.

Subjects will be recruited prospectively based on pre-specified enrollment criteria. Blood and urine samples will be collected after enrollment and at several timepoints, and various tests will be performed, including point-of-care L-FABP measurements on urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older on the day of the procedure
* Undergoing cardiac or vascular interventional procedures for diagnostic angiography, coronary intervention, TAVR or TAVI, with planned use of radiocontrast media within the next 30 days
* Able to provide informed consent
* Available to participate in follow-up visits
* eGFR < 45 within the last 90 days, or
* eGFR < 60 within the last 90 days with at least one (1) of the following risk factors:
* Diabetes
* Heart failure (acute or chronic)
* Anemia (hemoglobin < 12 g/dL for females and < 13 g/dL for males) within the last 90 days
* Age > 75 on the day of the procedure

Exclusion Criteria:

* Patient on dialysis or with eGFR < 15 within the last 30 days
* History of renal transplant
* Current use of immunosuppressive drugs other than prednisone < 10 mg/day
* Current clinically significant infection (including HIV, hepatitis)
* Presence of KDIGO Stage 1, 2, or 3 AKI within the last 7 days, according to KDIGO criteria
* Known or suspected nephritic or nephrotic syndrome.
* A current post-renal etiology of renal impairment
* Known allergy or hypersensitivity to radiographic contrast dye that cannot be pre-medicated
* Females that are known to be pregnant or nursing
* Participation within the last 30 days in another clinical trial involving use of any drug known to affect AKI and/or device known to affect AKI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients recruited from a healthcare setting that will be undergoing cardiac or vascular interventional procedures that are at elevated risk for developing AKI. At least 50% of the enrolled population will be undergoing an interventional procedure such as percutaneous coronary intervention (PCI), transcatheter aortic valve replacement (TAVR) or transcatheter aortic valve implantation (TAVI).
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of acute kidney injury | Within 2 days after a cardiac or vascular catheterization procedure involving the use of contrast media
  AKI defined as stage 1, 2, or 3 using the KDIGO criteria

CONTACTS AND LOCATIONS:
Overall Officials: Peter McCullough, Principal Investigator — Independent
Locations (6):
- United States (6):
  - Chandler Regional Medical Center, Chandler, Arizona
  - John Muir Health, Concord, California
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - University of Florida at Jacksonville, Jacksonville, Florida
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - University of Oklahoma, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noiri E, Doi K, Negishi K, Tanaka T, Hamasaki Y, Fujita T, Portilla D, Sugaya T. Urinary fatty acid-binding protein 1: an early predictive biomarker of kidney injury. Am J Physiol Renal Physiol. 2009 Apr;296(4):F669-79. doi: 10.1152/ajprenal.90513.2008. Epub 2008 Nov 19. PMID 19019918
- [Background] Yamamoto T, Noiri E, Ono Y, Doi K, Negishi K, Kamijo A, Kimura K, Fujita T, Kinukawa T, Taniguchi H, Nakamura K, Goto M, Shinozaki N, Ohshima S, Sugaya T. Renal L-type fatty acid--binding protein in acute ischemic injury. J Am Soc Nephrol. 2007 Nov;18(11):2894-902. doi: 10.1681/ASN.2007010097. Epub 2007 Oct 17. PMID 17942962
- [Background] Fujita D, Takahashi M, Doi K, Abe M, Tazaki J, Kiyosue A, Myojo M, Ando J, Fujita H, Noiri E, Sugaya T, Hirata Y, Komuro I. Response of urinary liver-type fatty acid-binding protein to contrast media administration has a potential to predict one-year renal outcome in patients with ischemic heart disease. Heart Vessels. 2015 May;30(3):296-303. doi: 10.1007/s00380-014-0484-9. Epub 2014 Feb 20. PMID 24554034
- [Background] Kamijo-Ikemori A, Hashimoto N, Sugaya T, Matsui K, Hisamichi M, Shibagaki Y, Miyake F, Kimura K. Elevation of urinary liver-type fatty acid binding protein after cardiac catheterization related to cardiovascular events. Int J Nephrol Renovasc Dis. 2015 Aug 18;8:91-9. doi: 10.2147/IJNRD.S88467. eCollection 2015. PMID 26316797
- [Background] Manabe K, Kamihata H, Motohiro M, Senoo T, Yoshida S, Iwasaka T. Urinary liver-type fatty acid-binding protein level as a predictive biomarker of contrast-induced acute kidney injury. Eur J Clin Invest. 2012 May;42(5):557-63. doi: 10.1111/j.1365-2362.2011.02620.x. Epub 2011 Nov 10. PMID 22070248
- [Background] Nakamura T, Sugaya T, Node K, Ueda Y, Koide H. Urinary excretion of liver-type fatty acid-binding protein in contrast medium-induced nephropathy. Am J Kidney Dis. 2006 Mar;47(3):439-44. doi: 10.1053/j.ajkd.2005.11.006. PMID 16490622